CLINICAL TRIAL: NCT02257047
Title: Red Yeast Rice and Subclinical Atherosclerosis in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chengdu PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yang Min, Ph.D, Chengdu PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RYR20140104
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Tea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RYR (Experimental): Patients under the treatment of red yeast rice
  Interventions: Dietary Supplement: RYR
- Control (Sham Comparator): Patients under the treatment of tea
  Interventions: Dietary Supplement: Tea

INTERVENTIONS:
Dietary Supplement: Tea
  Arms: Control
Dietary Supplement: RYR — red yeast rice
  Arms: RYR

SUMMARY:
To evaluate the effect of red yeast rice on subclinical atherosclerosis in patients with rheumatoid arthritis

ELIGIBILITY:
Inclusion Criteria:

* patients with a definite diagnose of rheumatoid arthritis(RA) were included if they met the classification criteria for RA established by the American Rheumatism Association (ACR) and European League Against Rheumatism (EULAR) in 2010
* aged from 18 to 75 years
* without conflict to the written, informed consent signed prior to the enrollment
* no severe hepatic or renal disorders
* no known carotid artery stenosis
* no coagulation disorders
* no hypertension

Exclusion Criteria:

* being in pregnancy, lactation period or under a pregnancy plan
* being allergic to the test drug
* not compatible for the trial medication
* without full legal capacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in Carotid intima-media thickness at 24 weeks | At 0 week, 12 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Chengdu Military Area Command PLA, Chengdu, Sichuan, China